CLINICAL TRIAL: NCT03956017
Title: Anti-oxidant Therapy and Postoperative Cardiac Events (ACE) Trial, Preoperative Intervention in Vascular Surgery
Acronym: ACE
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edward McFalls, CARDIOLOGIST, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND 119600 Coenzyme Q10
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Myocardial Injury
MeSH Terms: interventions — Ubiquinone; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ubiquinone (Experimental): Take oral tablets as directed (2x200 mg for 3 days prior to surgery)
  Interventions: Drug: Ubiquinone
- Placebo (Placebo Comparator): Take oral tablets as directed (2x200 mg for 3 days prior to surgery)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ubiquinone — Take oral tablets as directed (2x200 mg for 3 days prior to surgery)
  Other Names: CoQ10, Coenzyme Q10
  Arms: Ubiquinone
Drug: Placebo — Take oral tablets as directed (2x200 mg for 3 days prior to surgery)
  Other Names: Sugar pill, inactive substance
  Arms: Placebo

SUMMARY:
N Terminal (NT)-Pro b-type natriuretic peptide (BNP) levels provide incremental value in perioperative risk assessment prior to major non-cardiac surgery. The investigators will test whether pharmacologically lowering this biomarker with daily administration of CoQ10 for 3 days prior to elective vascular surgery will reduce adverse outcomes following the operation.

DETAILED DESCRIPTION:
Patients will be screened during their preoperative evaluation. Inclusion criteria include patients in need of an elective vascular operation. Exclusion criteria include urgent operation, known allergic reactions to CoQ10 and participation in another research study. Suitable participants will be randomly assigned to receive either CoQ10 (400 mg per day) versus Placebo for 3 days prior to surgery. A randomized, double blind trial will be used and a research pharmacist will guide the randomization process, blinded to clinical information. The primary end-point measures are BNP levels at 24 and 48 hours following the operation as well as the incidence of myocardial injury, defined by an elevated post-operative high-sensitivity troponin following high risk surgery. Secondary outcome measures include the magnitude of the troponin level, which is the change in the level compared with preoperative baseline troponin levels and adverse clinical cardiac outcomes during the hospitalization period, including death, non-fatal myocardial infarction, diagnosed by a cardiologist who is blinded to the treatment strategy and any coronary artery revascularization procedure. The study will be focused on 30-days following the vascular procedure but the investigators may plan to extend secondary outcome measures for 1 year post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* ELECTIVE HIGH RISK NON-CARDIAC SURGERY

Exclusion Criteria:

* REACTION TO COQ10

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 341 (Estimated)
Dates: Start 2013-08-05 (Actual); Primary Completion 2022-08-04 (Estimated); Study Completion 2022-08-04 (Estimated)

PRIMARY OUTCOMES:
BNP levels following surgery | 48 hours
  Peak values
Cardiac Troponin levels following surgery | 48 hours
  Peak values
Change in Troponin levels from baseline to peak | 48 hours
  Change from baseline to peak
Number of participants with adverse cardiac outcomes following surgery | 48 hours
  Myocardial Infarction (MI) and death

SECONDARY OUTCOMES:
Number of participants who died | 30 days
  All cause mortality
Number of participants requiring coronary revascularization | 30 days
  Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Grafting (CABG)
Number of participants with new heart failure | 30 days
  Heart failure, newly diagnosed by cardiologist
Number of participants with new onset Atrial Fibrillation (A-Fib) | 30 days
  New onset A-Fib
Number of participants with infection | 30 days
  Infection diagnosed by a primary care provider
Number of participants with a surgical graft failure | 30 days
  Primary surgical site graft failure
Length of stay | 30 days
  Length of stay in days for index hospitalization
Rate of readmission at 1 year following discharge | 1 year
  Any admission to hospital for 1 year post discharge

CONTACTS AND LOCATIONS:
Overall Officials: EDWARD MCFALLS, MD, Study Chair — SITE PI
Locations (1):
- Va Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Sharing plan will be left at the discretion of the VA funding organization and statistical site.

REFERENCES:
- [Derived] Khan A, Johnson DK, Carlson S, Hocum-Stone L, Kelly RF, Gravely AA, Mbai M, Green DL, Santilli S, Garcia S, Adabag S, McFalls EO. NT-Pro BNP Predicts Myocardial Injury Post-vascular Surgery and is Reduced with CoQ10: A Randomized Double-Blind Trial. Ann Vasc Surg. 2020 Apr;64:292-302. doi: 10.1016/j.avsg.2019.09.017. Epub 2019 Oct 17. PMID 31629852